CLINICAL TRIAL: NCT01918423
Title: The Effects of Lifestyle Intervention During Pregnancy in Obese Women on Offspring Adiposity and Metabolic Risk Factors- Comparison With Offspring of Normal Weight Women Not Participating in a Lifestyle Intervention Programme.
Brief Title: Lifestyle in Pregnancy and Offspring - Comparison Between Children Born to Obese Women and Children Born to Normal Weight Women
Acronym: LiPO
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mette Tanvig, Medical Doctor, Odense University Hospital
Other Study IDs: LiPO-2
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Childhood Obesity
Keywords: Childhood adiposity; Metabolic risk factors; Bone mineralization
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We have created a biobank of bloodsamples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Children of obese women from a RCT: Children born to obese women who were in the active intervention arm of the randomized controlled trial LiP. The lifestyle intervention during pregnancy consisted of two major components: dietary counseling and physical activity. Dietary counseling was performed by trained dieticians on four separate occasions at 15, 20, 28 and 35 weeks gestation.
  Interventions: Behavioral: Lifestyle intervention during pregnancy
- Children of obese mothers from a RCT, controls: Children born to obese mothers who were in the control arm of the randomized controlled trial LiP.
- Children born to normal weight women: Children born to women with a pregestationally normal BMI and who were not part of a lifestyle intervention programme during pregnancy.

INTERVENTIONS:
Behavioral: Lifestyle intervention during pregnancy — Energy requirements for each participants´ mother were individually estimated according to weight and level of activity during pregnancy. Women in the active intervention group were encouraged to be moderately physically active 30-60 minutes a day.Women in this group also had free full time membership in a fitness center for six months. In the fitness centers they had closed training classes with trained physiotherapists for one hour each week.
  Groups: Children of obese women from a RCT

SUMMARY:
Children born to obese women are at risk of increased adiposity and later adverse metabolic outcomes. We have conducted a follow-up study on an existing clinical trial, called the LiP study (Lifestyle in Pregnancy), registration number NCT00530439,in which 360 obese pregnant women were randomized to either lifestyle intervention or routine obstetric care. This present study follows the children until 3 years of age. We have the hypothesis, that the intervention during pregnancy results in a lower degree of adiposity and metabolic risk factors in the offspring. Clinical examination is taking place at age 2.5-3 years including anthropometric measurements, Dual energy x-ray (DXA) scans and blood samples measuring metabolic markers.In addition, we have included an extra control group of children born to normal weight women, who were not part of a lifestyle intervention program during pregnancy. We have the hypothesis that the children of the normal weight women have a better metabolic profile than the children born to the obese women.

ELIGIBILITY:
Inclusion Criteria:

- All children born to obese women who participated in the LiP study (a randomized controlled trial of lifestyle intervention during pregnancy) and children born at term to healthy women with a normal pregestational BMI.

Exclusion Criteria:

- The children born to normal weight women only: preterm birth, congenital anomalies, maternal gestational diabetes, maternal diabetes mellitus, severe medical conditions in either child or mother.

Ages: 30 Months to 40 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Three groups of children at the ages of 2.5 til 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Child body mass standard deviation score | On average 2.9 years of age

SECONDARY OUTCOMES:
anthropometric outcomes | On average 2.9 years of age
  Fat percent measured by DXA.

OTHER OUTCOMES:
Anthropometric and metabolic outcomes. Bone mineralization | On average 2.9 years of age
  BMI, Skinfold thicknesses, abdominal circumference, hip circumference, abdominal to hip circumference ratio, height, weight. DXA scan: fat mass, fat mass percent, lean mass, lean mass percent, body fat distribution. Bone mass density, bone mass content. Fasting blood glucose, HbA1C, fasting insulin, fasting c-peptide, fasting lipids; HDL; LDL, triglycerides, total cholesterol. 25-hydroxy vitamin D. Bone mineralization estimated with dual energy x-ray and a computer program estimating bone health index (BHI) from x-rays of the hand.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Tanvig, MD, Principal Investigator — Department of endocrinology, Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Jorgensen JS. The LiP (Lifestyle in Pregnancy) study: a randomized controlled trial of lifestyle intervention in 360 obese pregnant women. Diabetes Care. 2011 Dec;34(12):2502-7. doi: 10.2337/dc11-1150. Epub 2011 Oct 4. PMID 21972411
- [Derived] Tanvig M, Vinter CA, Jorgensen JS, Wehberg S, Ovesen PG, Beck-Nielsen H, Christesen HT, Jensen DM. Effects of lifestyle intervention in pregnancy and anthropometrics at birth on offspring metabolic profile at 2.8 years: results from the Lifestyle in Pregnancy and Offspring (LiPO) study. J Clin Endocrinol Metab. 2015 Jan;100(1):175-83. doi: 10.1210/jc.2014-2675. PMID 25343235
- [Derived] Tanvig M, Vinter CA, Jorgensen JS, Wehberg S, Ovesen PG, Lamont RF, Beck-Nielsen H, Christesen HT, Jensen DM. Anthropometrics and body composition by dual energy X-ray in children of obese women: a follow-up of a randomized controlled trial (the Lifestyle in Pregnancy and Offspring [LiPO] study). PLoS One. 2014 Feb 24;9(2):e89590. doi: 10.1371/journal.pone.0089590. eCollection 2014. PMID 24586896